CLINICAL TRIAL: NCT03548168
Title: Innovative Neurophysiological Techniques for Assessing Trunk Muscle Control and Function (iCAM)
Brief Title: Innovative Imaging of Cerebrum and Muscle (iCAM) Repeatability Study
Acronym: iCAM
Status: Completed | Type: Observational
Sponsor: Ohio University (Other)
Responsible Party: Sponsor
Other Study IDs: 17-F-23
Record Dates: First submitted 2018-05-24; First posted 2018-06-07 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-02

CONDITIONS: Low Back Pain; Aging
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Healthy Adults: Eligible healthy young adults, aged 18-30 years, will participate in testing experiments to test-retest reliability of the muscle functional magnetic resonance imaging (mfMRI) and functional magnetic resonance imaging (fMRI) techniques that were developed in order to study the neural control of trunk muscles.
- Low Back Pain: Eligible young adults, aged 18-30 years, with chronic low back pain will participate in testing experiments to test-retest reliability of the muscle functional magnetic resonance imaging (mfMRI) and functional magnetic resonance imaging (fMRI) techniques that were developed in order to study the neural control of trunk muscles.
- Older Adults: Eligible healthy middle aged and older adults, aged 55 years and older, will participate in testing experiments to test-retest reliability of the muscle functional magnetic resonance imaging (mfMRI) and functional magnetic resonance imaging (fMRI) techniques that were developed in order to study the neural control of trunk muscles.
- Trunk Experts: Eligible healthy middle aged and older adults, aged 55 years and older, with high levels of trunk muscle control (ie. individuals with expertise in the Pilates Method of exercise) will participate in testing experiments to test-retest reliability of the muscle functional magnetic resonance imaging (mfMRI) and functional magnetic resonance imaging (fMRI) techniques that were developed in order to study the neural control of trunk muscles.

SUMMARY:
Impairments in postural control are linked to low back pain and reductions in physical function in the elderly. Unfortunately, many techniques to assess the neural control of movement are not feasible, or directly applicable, to the trunk musculature. In a prior pilot study, we developed and optimized innovative approaches to study these muscles. We will continue to develop a reliable, fMRI protocol that investigates the activity of the motor cortical networks of selected trunk muscles (specific aim 1). We will also continue the development a reliable muscle functional MRI (mfMRI) protocol to assess the spatial muscle activation patterns of the deeper lumbopelvic muscles (specific aim 2). We will examine the test-retest reliability of these approaches in four distinct target populations: healthy adults, adults with chronic low back pain, older adults, and older adults with high levels of trunk muscle control (i.e., individuals with expertise in Pilates). By enrolling groups of various levels of trunk muscle control, pathology state and age, we will be able to not only determine the intra-individual reliability, but also the inter-individual reliability as we expect the variability of the measures to be influenced by physical ability, pain state and age. Lastly, in an exploratory aim we will examine the association of our novel neurophysiological measures from Aim 1 and 2 with classic biomechanical and muscle function measures (e.g., trunk extensor strength and trunk extensor steadiness). Successfully developing reliable techniques of this nature will result in new and improved research tools for conducting rigorous studies of therapeutic approaches, such as spinal manipulation and yoga, within the context of trunk muscle control and function.

DETAILED DESCRIPTION:
Impairments in postural control are linked to low back pain and reductions in physical function in the elderly. Unfortunately, many techniques to assess the neural control of movement are not feasible or directly applicable to the trunk musculature. We have developed an innovative approach to study these muscles. Further development of these techniques will have applicability for the study of the physiological effects and mechanisms of many complementary and integrative health practices (e.g., mind and body approaches). Many of these approaches are used to target back pain (e.g., spinal manipulation, acupuncture) and/or involve therapeutic strategies that have a large focus on postural control (e.g., yoga, Tai Chi). Thus, developing novel and reliable techniques to study the neural control of the trunk muscles will have broad impact to the complementary and integrative health field.

Specific Aim 1. To develop a reliable neurophysiological technique to examine activity of the motor neural networks of selected trunk muscles. Approach: We have previously conducted pilot testing exploring the feasibility of obtaining high quality MRI data with various standardized trunk tasks and biofeedback variations. Once we identified the most promising tasks and MRI compatible data collection techniques, we conducted an optimization study in order to ascertain which method of task performance resulted in the highest level of image quality. We will now conduct a test-retest reliability experiment to determine the reproducibility of our targeted outcome measures. We will focus our reliability analysis on the bilateral primary sensorimotor cortex (Brodmann area 4a, 4b, 1, 2, 3a and 3b) and premotor cortex (Brodmann area 6). In addition, contrasts between two testing sessions will be completed to determine if any brain regions activated significantly more or less between sessions.

Specific Aim 2. To develop a reliable neurophysiological technique to examine spatial muscle activity of selected lumbopelvic musculature (e.g., psoas, iliacus, multifidus, erector spinae, quadratus lumborum). Approach: We have conducted pilot testing that explored the feasibility of obtaining high quality MRI data of various muscles under resting conditions as well as following different standardized tasks. We first identified the most promising muscles to evaluate and then explored which tasks (or tasks sequences) resulted in increased transverse relaxation times (T2) of these muscles. We refined our pulse sequence protocol to optimize our ability to detect an increase in T2 associated with task performance. We will now conduct a test-retest reliability experiment to determine the reproducibility of the primary outcome measures of interest (resting T2 and percent increase in T2 following task performance).

Exploratory Specific Aim 3. To examine the association of the novel neurophysiological measures from Aim 1 and 2 with classic biomechanical and muscle function measures (e.g., trunk extensor strength, trunk extensor force-matching steadiness). The neurophysiological assessments developed as a part of Aim 1 and 2 provide unique information regarding the mechanisms of motor control related to trunk musculature that have typically been very difficult to quantify. This mechanistic approach is bolstered by the ability to correlate the underlying neurophysiology of trunk function with the more traditional clinical measures of performance. Such an approach bolsters the translational capability of this investigation as the neurophysiology of low-cost clinical measures are established in addition to the development of novel intervention outcome tools.

Study Participants: Up to 50 individuals will participate in the reliability experiments. To increase the generalizability of our findings and allow for preliminary data for effect size estimates for future work, we will enroll four cohorts of study participants: healthy young adults, young adults with chronic low back pain, healthy older adults and healthy older adults with expertise in trunk muscle control (i.e., individuals with expertise in Pilates).

Expected Outcomes: We anticipate being able to demonstrate test-retest reliability utilizing two newly developed neurophysiological imaging techniques that will permit 1) examination of the activity of the motor cortical networks during an active trunk task, and 2) examination of muscle activation patterns of small and deep trunk extensor muscles that are very difficult, if not impossible, to study with more classical techniques such as electromyography. Our goal is to demonstrate an association with outcomes of these new imaging techniques with more classic neurophysiological motor outcomes for broad applicability to numerous patient populations that we believe, in the long term, will advance our understanding of trunk muscle control and function.

In this application we propose to perform the test- retest reliability experiments for the fMRI and mfMRI techniques that were previously developed in the pilot testing.

ELIGIBILITY:
1. Healthy young adults Eligible subjects are males and females aged 18-30 years with no significant health issues

   Inclusion Criteria:

   A subject must meet the following criteria to be eligible for inclusion in the study:
   * Men and women aged 18- 30 years, with no significant health issues or conditions that, in the investigator's opinion, would limit the subject's ability to complete the study activities or that would impact the capability to get an accurate measurement of study endpoints.
   * Body mass index (BMI) between 17 and 30 kg/m2.
   * Willing to undergo multiple MRI sessions.
   * Willing and able to return for all visits and complete all study-related activities.
   * Able to read, understand, and complete study-related questionnaires
   * Able to read and understand, and willing to sign the informed consent form (ICF).

   Exclusion criteria:

   A subject who meets any of the following criteria will be excluded from the study:
   * Having body dimensions that exceed the MRI or exercise equipment limits.
   * Unable to undergo MRI (e. g. body containing any metallic medical devices or equipment, including heart pacemakers, metal prostheses, implants or surgical clips, any prior injury from shrapnel or grinding metal, exposure to metallic dusts, metallic shavings or having tattoos containing metallic dyes)
   * Abnormal or uncontrolled blood pressure at the screening visit defined as BP > 180/100 mmHg.
   * Positive pregnancy test.
   * Having a personal history of the following neurological disorders: Alzheimers, Amyotrophic Lateral Sclerosis, Multiple Sclerosis, Parkinsons, Stroke
   * Having a personal history of the following cardiorespiratory disorders: Congestive heart failure, Heart attack in past 24 months
   * Having a personal history of the following musculoskeletal disorders: Rheumatoid Arthritis, pathologic fractures of the spine, avascular necrosis or osteonecrosis, severe osteoarthritis. Including a history of spine surgery or a hip arthroplasty.
   * Having neurological symptoms (ie. burning, numbness, tingling sensations into the legs), muscle weakness associated with neural dysfunction (i.e. foot drop), or episodes of incontinence of bowel or bladder.
   * Having active cancer
   * Blindness
   * Having used opioids or muscle relaxants within 30 days prior to study enrollment.
   * Reports being pregnant, lactating, or that they anticipate becoming pregnant in the next 3-months. If a woman becomes pregnant while on study protocol they will be withdrawn from the study.
   * Reports unexplained weight loss over the past month (greater than 10 lbs).
   * Failure to provide informed consent.
2. Young adults with chronic low back pain (CLBP) Eligible subjects are males and females aged 18- 30 years with no significant health issues except self report of CLBP

   Inclusion Criteria:

   A subject must meet the following criteria to be eligible for inclusion in the study:
   * Men and women aged 18- 30 years, with no significant health issues or conditions that, in the investigator's opinion, would limit the subject's ability to complete the study activities or that would impact the capability to get an accurate measurement of study endpoints.
   * Body mass index (BMI) between 17 and 30 kg/m2.
   * Willing to undergo multiple MRI sessions.
   * Willing and able to return for all visits and complete all study-related activities.
   * Able to read, understand, and complete study-related questionnaires.
   * Able to read and understand, and willing to sign the informed consent form (ICF).
   * Reports average pain intensity (assessed using the Numerical Pain Rating (NPRS) scale) over the past week greater than or equal to 3 on a 0-10 numerical pain scale.
   * Oswestry Low Back Pain Disability Questionnaire score > 20% (moderate disability and above).
   * Answers yes to the following questions:

   Have you had low back pain constantly or on most days for the last three months? Has your back pain caused you to seek care or consultation from a health care provider?

   Exclusion criteria:

   A subject who meets any of the following criteria will be excluded from the study:
   * Having body dimensions that exceed the MRI or exercise equipment limits.
   * Unable to undergo MRI (e. g. body containing any metallic medical devices or equipment, including heart pacemakers, metal prostheses, implants or surgical clips, any prior injury from shrapnel or grinding metal, exposure to metallic dusts, metallic shavings or having tattoos containing metallic dyes)
   * Abnormal or uncontrolled blood pressure at the screening visit defined as BP > 180/100 mmHg.
   * Positive pregnancy test.
   * Having a personal history of the following neurological disorders: Alzheimers, Amyotrophic Lateral Sclerosis, Multiple Sclerosis, Parkinsons, Stroke
   * Having a personal history of the following cardiorespiratory disorders: Congestive heart failure, Heart attack in past 24 months
   * Having a personal history of the following musculoskeletal disorders: Rheumatoid Arthritis, pathologic fractures of the spine, avascular necrosis or osteonecrosis, severe osteoarthritis. Including a history of spine surgery or a hip arthroplasty
   * Having neurological symptoms (ie. burning, numbness, tingling sensations into the legs), muscle weakness associated with neural dysfunction (i.e. foot drop), or episodes of incontinence of bowel or bladder
   * Having active cancer
   * Blindness
   * Having used opioids or muscle relaxants within 30 days prior to study enrollment.
   * Reports being pregnant, lactating, or that they anticipate becoming pregnant in the next 3-months. If a woman becomes pregnant while on study protocol they will be withdrawn from the study.
   * Reports unexplained weight loss over the past month (greater than 10 lbs).
   * Reports having pending litigation related to an episode of LBP or are receiving any type of disability services related to low back pain.
   * Reports having received any manual therapy intervention applied to the spine 30 days prior to first study intervention.
   * Reports current drug or alcohol use or dependence that, in the opinion of the PIs, would interfere with adherence to study requirements.
   * Failure to provide informed consent.
3. Healthy middle-aged and older adults Eligible subjects are males and females aged 55+ years with no significant health issues

   Inclusion Criteria:

   A subject must meet the following criteria to be eligible for inclusion in the study:
   * Men and women over 55 years of age, with no significant health issues or conditions that, in the investigator's opinion, would limit the subject's ability to complete the study activities or that would impact the capability to get an accurate measurement of study endpoints.
   * Body mass index (BMI) between 17 and 30 kg/m2.
   * Willing to undergo multiple MRI sessions.
   * Willing and able to return for all visits and complete all study-related activities.
   * Able to read, understand, and complete study-related questionnaires
   * Able to read and understand, and willing to sign the informed consent form (ICF).

   Exclusion criteria:

   A subject who meets any of the following criteria will be excluded from the study:
   * Having body dimensions that exceed the MRI or exercise equipment limits.
   * Unable to undergo MRI (e. g. body containing any metallic medical devices or equipment, including heart pacemakers, metal prostheses, implants or surgical clips, any prior injury from shrapnel or grinding metal, exposure to metallic dusts, metallic shavings or having tattoos containing metallic dyes)
   * Abnormal or uncontrolled blood pressure at the screening visit defined as BP > 180/100 mmHg.
   * Positive pregnancy test.
   * Having a personal history of the following neurological disorders: Alzheimers, Amyotrophic Lateral Sclerosis, Multiple Sclerosis, Parkinsons, Stroke
   * Having a personal history of the following cardiorespiratory disorders: Congestive heart failure, Heart attack in past 24 months
   * Having a personal history of the following musculoskeletal disorders: Rheumatoid Arthritis, pathologic fractures of the spine, avascular necrosis or osteonecrosis, severe osteoarthritis. Including a history of spine surgery or a hip arthroplasty
   * Having neurological symptoms (ie. burning, numbness, tingling sensations into the legs), muscle weakness associated with neural dysfunction (i.e. foot drop), or episodes of incontinence of bowel or bladder
   * Having active cancer
   * Blindness
   * Having used opioids or muscle relaxants within 30 days prior to study enrollment.
   * Reports being pregnant, lactating, or that they anticipate becoming pregnant in the next 3-months. If a woman becomes pregnant while on study protocol they will be withdrawn from the study.
   * Reports unexplained weight loss over the past month (greater than 10 lbs).
   * Failure to provide informed consent.
4. Healthy middle-aged and older adults with high levels of trunk muscle control (ie. individuals with expertise in the Pilates Method of exercise)

Eligible subjects are males and females aged 55+ years with no significant health issues

Inclusion Criteria:

A subject must meet the following criteria to be eligible for inclusion in the study:

* Men and women over 55 years of age, with no significant health issues or conditions that, in the investigator's opinion, would limit the subject's ability to complete the study activities or that would impact the capability to get an accurate measurement of study endpoints.
* Reports being trained in the Pilates method exercises and has been performing these exercises 2 times per week for the past one year.
* Body mass index (BMI) between 17 and 30 kg/m2.
* Willing to undergo multiple MRI sessions.
* Willing and able to return for all visits and complete all study-related activities.
* Able to read, understand, and complete study-related questionnaires
* Able to read and understand, and willing to sign the informed consent form (ICF).

Exclusion criteria:

A subject who meets any of the following criteria will be excluded from the study:

* Having body dimensions that exceed the MRI or exercise equipment limits.
* Unable to undergo MRI (e. g. body containing any metallic medical devices or equipment, including heart pacemakers, metal prostheses, implants or surgical clips, any prior injury from shrapnel or grinding metal, exposure to metallic dusts, metallic shavings or having tattoos containing metallic dyes)
* Abnormal or uncontrolled blood pressure at the screening visit defined as BP > 180/100 mmHg.
* Positive pregnancy test.
* Having a personal history of the following neurological disorders: Alzheimers, Amyotrophic Lateral Sclerosis, Multiple Sclerosis, Parkinsons, Stroke
* Having a personal history of the following cardiorespiratory disorders: Congestive heart failure, Heart attack in past 24 months
* Having a personal history of the following musculoskeletal disorders: Rheumatoid Arthritis, pathologic fractures of the spine, avascular necrosis or osteonecrosis, severe osteoarthritis. Including a history of spine surgery or a hip arthroplasty
* Having neurological symptoms (ie. burning, numbness, tingling sensations into the legs), muscle weakness associated with neural dysfunction (i.e. foot drop), or episodes of incontinence of bowel or bladderHaving active cancer
* Blindness
* Having used opioids or muscle relaxants within 30 days prior to study enrollment.
* Reports being pregnant, lactating, or that they anticipate becoming pregnant in the next 3-months. If a woman becomes pregnant while on study protocol they will be withdrawn from the study.
* Reports unexplained weight loss over the past month (greater than 10 lbs).
* Failure to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Young healthy adults, young healthy adults with chronic low back pain, healthy middle aged/older adults, and health middle aged/older adults with high levels of trunk muscle control.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2018-05-18 (Actual); Primary Completion 2020-05-03 (Actual); Study Completion 2020-05-05 (Actual)

PRIMARY OUTCOMES:
Trunk extensor fMRI signal intensity | 3 years
  Physiological measure of brain efficiency in activating the trunk muscles

CONTACTS AND LOCATIONS:
Overall Officials: Brian Clark, PhD, Principal Investigator — Ohio Musculoskeletal and Neurological Institute
Locations (1):
- Ohio Musculoskeletal and Neurological Institute (OMNI) at Ohio University, Athens, Ohio, United States

IPD SHARING:
Plan to Share IPD: No